CLINICAL TRIAL: NCT00582244
Title: Cognitive Behavioral Therapy (CBT) and Physical Exercise for Climacteric Symptoms in Breast Cancer Patients Experiencing Treatment-Induced Menopause: a Multicenter Randomized Trial
Acronym: EVA project
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Prof. dr. N.K. Aaronson, NKI-AVL
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NKI 2006-3470; NKI 2006-3470
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Menopausal Symptoms in Breast Cancer Patients With Treatment-Induced Complaints
Keywords: Menopausal symptoms; Quality of Life; Breast cancer; Multicenter trial
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): CBT and relaxation.
  Interventions: Behavioral: CBT and relaxation
- 2 (Experimental): Physical activity
  Interventions: Behavioral: Physical activity
- 3 (Experimental): CBT and physical activity
  Interventions: Behavioral: CBT and physical activity
- 4 (No Intervention): Control group
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: CBT and relaxation — Group A: CBT and relaxation.
  Arms: 1
Behavioral: Physical activity — Group B: Physical exercise program.
  Arms: 2
Behavioral: CBT and physical activity — Group AB: Combined CBT and exercise program. Women assigned to Group AB will undergo the CBT and exercise elements of the program concurrently. To as great an extent as possible, the on-site CBT and in-clinic exercise training sessions will be scheduled on the same day.
  Arms: 3
Other: Control group — Waiting list control group
  Arms: 4

SUMMARY:
Background: Breast cancer is the most common form of cancer among women in the Netherlands. Approximately 11,000 women are diagnosed with breast cancer annually, of whom about 30% are below 50 years of age. Premenopausal women with breast cancer treated with chemotherapy or hormonal therapy may experience a premature onset of the menopause. Estrogen deficiency following adjuvant treatments leads to primary endocrine symptoms, including vasomotor and urogenital problems. Secondary symptoms include insomnia due to night sweats, dyspareunia due to vaginal dryness, weight gain, and psychological distress. The symptoms resulting from accelerated estrogen withdrawal can be pronounced and severe, and may adversely affect women's sexual functioning, body image, and overall HRQL. Healthy women who enter natural menopause are often prescribed hormone replacement therapy (HRT) to alleviate vasomotor and sexual symptoms. However, due to possible tumor-promoting effects, HRT is contraindicated for patients with a history of breast cancer. For these women, non-hormonal medications are frequently prescribed to treat vasomotor symptoms. Although these medications have been shown to yield moderate symptom relief, they also have a number of bothersome side effects. To alleviate urogenital symptoms, local vaginal moisturizing or estrogen cream is often prescribed. There is growing evidence that cognitive behavioral therapy (CBT) including relaxation techniques, and physical exercise may effectively reduce vasomotor symptoms in naturally occurring menopause. CBT and relaxation techniques are aimed primarily at the modification of precipitants of hot flushes and at stress management. Physical exercise on a regular basis affects neurotransmitters, which regulate central thermoregulation.

Purpose: The proposed study will evaluate the efficacy of a supportive intervention program in alleviating menopausal symptoms, improving sexual functioning and enhancing the quality of life of younger women (< 50 years) with breast cancer who have become prematurely menopausal as a result of their treatment. Specifically, the study will evaluate CBT including relaxation (A), physical exercise (B), and a combination of A and B.

Plan of investigation: This multicenter study will employ a prospective, full-factorial design. In total, 325 consenting women will be randomized to group A, group B, group AB or a usual care, 'waiting list' control group (N = 81-81 per group). Upon completion of the study, the patients assigned to the control group will be given the opportunity to undergo either the A or B intervention program. The program will begin with a structured assessment of the target symptoms: hot flushes, night sweating and vaginal dryness. The overriding goal of the intervention is to provide symptomatic women with information skills and support to manage their symptoms more effectively. For group A, the intervention will consist of 6 weekly group CBT sessions of 1.5 hours, of 15 minutes of daily homework and a booster session at 3 months. The CBT will focus on understanding and self-control of menopausal symptoms. Relaxation techniques (paced respiration and muscle relaxation) will focus on the reduction of sympathetic nervous system activity, and are expected to have a positive impact on the frequency and intensity of hot flushes. For group B, the intervention will be an individually tailored, 12 week home-based physical exercise program of 2.5-3 hours per week, with instructions provided in-clinic on 2 occasions, and telephone support on 2 additional, interim occasions. The physical exercise program is intended to enhance fitness levels, in general, and to improve thermoregulation specifically related to hot flushes. Group AB will receive both the CBT and exercise program elements. Women allocated to the intervention groups will be asked to complete a battery of questionnaires assessing menopausal symptoms (the primary outcome), sexuality, body- and self-image, psychological distress and generic HRQL prior to the start of the program (baseline, T0), at 12 weeks (T1) and at 6 months follow-up (T2). Women allocated to the control group will complete the same questionnaire battery at parallel points in time.

Results/ relevance: If demonstrated to be effective, the availability of a structured supportive intervention program (modules A, B or AB) will be a welcome addition to regular medical care offered to breast cancer patients with treatment-induced menopause. It is anticipated that such a program will have direct benefit in terms of symptoms relief and the improvement of patients' HRQL.

ELIGIBILITY:
Inclusion Criteria:

The study sample will be composed of 325 women, younger than 50 years of age, with histologically confirmed primary breast cancer (stages: T1 - T4, N0 - N1 and M0). All women will have been premenopausal at the time of diagnosis, have completed adjuvant chemotherapy (with the exception of herceptin, which can continue to receive) a minimum of 4 months and a maximum of 5 years prior to study entry. Women may currently be receiving adjuvant hormonal therapy. All women should be disease-free at time of study entry. Potentially eligible women will be screened for the presence of at least one of the following 3 menopausal symptoms during the previous 2-month period: hot flushes, sweating and/or vaginal dryness.

Exclusion Criteria:

Women will be excluded from the study if they lack basic proficiency in Dutch, if they have serious cognitive or psychiatric problems, or serious physical comorbidity that would preclude them from participating in a physical exercise program. Since physical exercise may be contraindicated as a treatment for hot flushes in obese women, 49 patients with a BMI ≥ 30 will be excluded from the study. Patients participating in concurrent studies or rehabilitation programs containing psychosocial interventions will also be excluded.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 325 (Estimated)
Dates: Start 2008-01; Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Menopausal symptoms | 6 months

SECONDARY OUTCOMES:
Vasomotor symptoms; urinary symptoms; sexuality; body- and self image; psychological distress; quality of life | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Neil Aaronson, Prof, Principal Investigator — NKI-AvL

REFERENCES:
- [Derived] Duijts SF, van Beurden M, Oldenburg HS, Hunter MS, Kieffer JM, Stuiver MM, Gerritsma MA, Menke-Pluymers MB, Plaisier PW, Rijna H, Lopes Cardozo AM, Timmers G, van der Meij S, van der Veen H, Bijker N, de Widt-Levert LM, Geenen MM, Heuff G, van Dulken EJ, Boven E, Aaronson NK. Efficacy of cognitive behavioral therapy and physical exercise in alleviating treatment-induced menopausal symptoms in patients with breast cancer: results of a randomized, controlled, multicenter trial. J Clin Oncol. 2012 Nov 20;30(33):4124-33. doi: 10.1200/JCO.2012.41.8525. Epub 2012 Oct 8. PMID 23045575
- [Derived] Duijts SF, Oldenburg HS, van Beurden M, Aaronson NK. Cognitive behavioral therapy and physical exercise for climacteric symptoms in breast cancer patients experiencing treatment-induced menopause: design of a multicenter trial. BMC Womens Health. 2009 Jun 6;9:15. doi: 10.1186/1472-6874-9-15. PMID 19500403